CLINICAL TRIAL: NCT03750396
Title: Local Treatment in Addition to Endocrine Therapy in ER-positive/HER2-negative Oligo-metastatic Breast Cancer (CLEAR): a Multicentre, Single -Arm, Phase 2 Trial
Brief Title: Local Treatment in ER-positive/HER2-negative Oligo-metastatic Breast Cancer
Acronym: CLEAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Collaborators: Severance Hospital (Other); Samsung Medical Center (Other); Asan Medical Center (Other)
Responsible Party: Principal Investigator, Joon Jeong, Professor, Gangnam Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEAR
Record Dates: First submitted 2018-11-16; First posted 2018-11-23 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Breast Cancer; Recurrent Breast Cancer; Stereotactic Body Radiotherapy; Estrogen Receptor Positive Tumor; Her2-negative Tumor; Surgery
Keywords: Oligometastasis; Local treatments
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiosurgery; Radiofrequency Ablation

STUDY DESIGN:
Intervention Model Description: Endocrine therapy is a standard-of-care for 1st line treatment in the patients with ER+/HER2- metastatic breast cancer.
  Local treatments for metastatic lesions will be added in this group.
  All patients will undergo local treatments in addition to endocrine therapies.
  Local treatments include modalities described below:
  i) Surgical resection: the achievement of tumor-free margin is not obligatory.
  ii) Stereotactic body radiotherapy
  iii) Radiofrequency ablation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endocrine and local treatments (Experimental): Endocrine therapy is a standard-of-care for 1st line treatment in the patients with ER+/HER2- metastatic breast cancer.
  Endocrine options included aromatase inhibitors, aromatase inhibitors with CDK4/6 inhibitors, fulvestrant, fulvestrant with CDK4/6 inhibitors, everolimus with exemestane, tamoxifen. For premenopausal women, agents for ovarian function suppression using GnRH agonists or surgical ovarian ablation including bilateral salpingo-oophorectomy are allowed.
  Local treatments for metastatic lesions will be added in this group.
  Local treatments include modalities described below:
  i) Surgical resection: the achievement of tumor-free margin is not obligatory. ii) Stereotactic body radiotherapy iii) Radiofrequency ablation
  Interventions: Procedure: Surgical resection; Radiation: Stereotactic body radiotherapy; Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Surgical resection — Surgical resection for their metastatic lesions will be performed. Achievement of tumor-free margin is not mandatory.
Radiation: Stereotactic body radiotherapy — Deliver appropriate metastasis directed radiotherapy while minimizing exposure of surrounding normal tissues. Total radiation dose and fractions are various according to metastatic lesions (57~97.5Gy/6~10 Fraction).
  Other Names: SBRT
Procedure: Radiofrequency ablation — RFA is a localized thermal treatment technique designed to induce tumor destruction by heating the tumor tissue to temperatures that exceed 60℃. The alternating current of radiofrequency waves passing down from an uninsulated electrode tip into the surrounding tissues generates changes in the direction of ions and creates ionic agitation and frictional heating. This tissue heating then drives extracellular and intracellular water out of the tissue, resulting in tissue destruction by coagulative necrosis.
  Other Names: RFA

SUMMARY:
Local treatment in addition to endocrine treatment as 1st line for oligo-metastatic ER-positive/HER2-negative breast cancer.

DETAILED DESCRIPTION:
Local treatment included surgical resection, stereotactic body radiotherapy, palliative radiotherapy, and radiofrequency ablation. Stereotactic body radiotherapy is preferred as a radiation modality.

Endocrine therapies with/without target therapy including CDK4/6 inhibitors or mTOR inhibitors are the mainstay of 1st line treatment for ER-positive/HER2-negative metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

-ER-positive/HER2-negative in primary tumor

* Oligometastases: ≤ 2 lesions in single organ or site (lung, bone, liver, adrenal glands, distant LNs)
* Recurrent cancer after completion of primary treatment (RFI≥1year)
* Metastatic lesions are feasible for resection or radiotherapy (Size≤3cm)

Exclusion Criteria:

* De Novo metastatic cancer at initial diganosis
* Recurrence-free inverval < 1 year

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically woman
Enrollment: 110 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From the date of registration to the date of first PFS failure or last follow-up; assessed up to 6 years; Median PFS of all registered patients will be over 30 months
  Failure: progression or death due to any cause

SECONDARY OUTCOMES:
Overall survival | From the date of registration to the date of death or last follow-up; assessed up to 10 years
  Failure: death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Joon Jeong, Ph.D., Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea